CLINICAL TRIAL: NCT01703117
Title: Glutamatergic Dysfunction in Cognitive Aging: Riluzole in Mild Alzheimer's Disease
Brief Title: Riluzole in Mild Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Principal Investigator, Ana Pereira, Principal Investigator; Assistant Professor of Neurology and Neuroscience, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 18-0623; APE-0792 (Other: Rockefeller University)
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- age matched cohort 50-95 years old (Experimental): 20-22 subjects between the ages of 50-95 will receive riluzole
  Interventions: Drug: Riluzole
- 24 subjects between 50-95 years old (Placebo Comparator): 20-22 subjects between 50-95 will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — 20-22 subjects between the ages of 60-85 will receive study drug.
  Other Names: no other names
  Arms: age matched cohort 50-95 years old
Drug: Placebo — 20-22 subjects between the ages of 60-85 will receive placebo
  Other Names: no other names
  Arms: 24 subjects between 50-95 years old

SUMMARY:
Cognitive aging is a major source of disability in an increasingly aging population. The paucity of effective treatments for cognitive aging disorders, and most importantly in Alzheimer's disease instigates a need for further research into novel therapeutic possibilities. Alzheimer's disease is the most common neurodegenerative disorder and its prevalence steeply increases. Glutamate-mediated excitotoxicity in neuropsychiatric disorders and in particular in Alzheimer's disease has been shown to cause significant cerebral damage. Early effective therapeutic intervention in Alzheimer's disease is critical in order to prevent or at least slow down neuropathological progression that will lead to widespread irreversible neuronal loss and significant cognitive dysfunction. Riluzole, a glutamate modulator agent, will be tested in mild Alzheimer's disease patients. Cognitive functional changes along with two established in vivo biomarkers, namely, Magnetic Resonance Spectroscopy (MRS) and Fluorodeoxyglucose (18F) positron emission tomography (FDG-PET) will be evaluated.

DETAILED DESCRIPTION:
A double-blinded, randomized, placebo-controlled study will be performed. Forty-two individuals with a diagnosis of mild Alzheimer's disease between 50-95 years old will complete the study. All forty-two individuals will have been on an acetylcholinesterase inhibitor, which is FDA approved for the treatment of Alzheimer's disease, for at least 2 months prior to initiating the study, unless the medication was not previously tolerated. Twenty to twenty-two mild Alzheimer's disease patients will receive riluzole and another 20-22 will receive a placebo. All patients will have a neurological evaluation and neuropsychological tests performed to confirm that they meet criteria for probable Alzheimer's disease set out by the National Institute on Aging - Alzheimer's disease Association that recently revisited the NINCDS-ADRDA criteria along with FDG-PET biomarker consistent with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; 50 - 95 years old with mild Alzheimer's disease determined after neurological and neuropsychological evaluation following the National Institute on Aging - Alzheimer's disease Association criteria that recently revisited the NINCDS-ADRDA criteria. For mild Alzheimer's disease, Clinical Dementia Ratings Scale (CDR) should be 0.5 or 1 and Mini Mental State Examination (MMSS) between 19 and 27.
* Must be on donepezil (Aricept®) or rivastigmine (Exelon®) or galantamine (Razadyne®) at a consistent dose for at least 2 months. Patients will be considered for inclusion if they were previously unable to tolerate acetylcholinesterase inhibitors and as a result, are no longer on the medication for at least 2 months.
* Must be fluent in English
* The subject will appoint or have previously appointed a health care proxy specifically designated for research consent and that this be documented.

Exclusion Criteria:

* Severe Alzheimer's disease and other dementias as determined by neuropsychological testing and neurological evaluation.
* Previous riluzole treatment.
* MRI contraindication (severe claustrophobia, metal implants, shunts, pacemaker, joint implants, metal valves).
* Currently taking medications that either have evidence of glutamatergic activity or has previous MRS evidence of effects on brain glutamate levels at the discretion of the PI such as memantine, lamotrigine, lithium, opiates, bupropion, psychostimulants such as amphetamines and methylphenidate, tricyclic antidepressants, benzodiazepines and any other drug that the investigators judge might interfere with the study. (subjects on those medications may still be included in the study however only the values of NAA from MRS will be utilized and not the glutamate measurements).
* Currently a user of the following illicit drugs: cocaine, methylenedioxymethamphetamine (MDMA) ("ecstasy"), heroin and other opioids or has a history of drug or alcohol abuse within the past 5 years.
* Serum creatinine >1.5 times the upper limit of normal.
* Abnormal liver function test (greater than 2 times the upper limit of normal for alanine aminotransferase (ALT) or aspartate aminotransferase (AST); or bilirubin >1.5 times the upper limit of normal.
* History of brain disease including Parkinson's Disease, severe brain trauma, seizures, history of stroke, clinically significant lacunar infarct in a region important for cognition or multiple lacunes or a cortical infarct or focal lesions of clinical significance, multiple sclerosis, mental retardation, normal pressure hydrocephalus, central nervous system (CNS) tumor, Huntington's disease, subdural hematoma or other serious neurological disorder.
* Uncontrolled diabetes mellitus (Hba1c higher than 7) or chronically uncontrolled hypertension.
* Subject must not be taking Namenda® (memantine) for 6-weeks prior to study entrance.
* Currently taking any concomitant hepatotoxic drugs such as allopurinol, methyldopa and sulfasalazine.
* Any unstable serious co-existing medical condition(s) including but not limited to myocardial infarction, coronary artery disease requiring coronary bypass surgery, unstable angina, clinically evident congestive heart failure within 6 months prior to the screening visit.
* Current smoker or user of nicotine-containing products, such as chewing tobacco, nicotine patch or gum for the past 2 months.
* Current untreated major depression defined by Geriatric Depression Scale > 20.
* Participation in any investigational or marketed drug or device trial within 30 days prior to the screening visit.
* Significant neuropsychiatric illnesses such as bipolar disorder, schizophrenia, moderate-severe anxiety, vascular dementia, Creutzfeldt-Jakob dementia, HIV dementia, and dementia in other specified diseases.
* Subjects who have been on donepezil for longer than 5 years.
* Weight> 300 pounds.
* Lactose intolerance.
* Any medical or social condition that, in the opinion of the Investigator, might pose additional risk to the participant or confound the results of the study.
* Positive Hepatitis Serology (Hep. B antigen+ or Hep. C antibody+)

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Pereira, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Rockefeller University, New York, New York

REFERENCES:
- [Result] Matthews DC, Mao X, Dowd K, Tsakanikas D, Jiang CS, Meuser C, Andrews RD, Lukic AS, Lee J, Hampilos N, Shafiian N, Sano M, David Mozley P, Fillit H, McEwen BS, Shungu DC, Pereira AC. Riluzole, a glutamate modulator, slows cerebral glucose metabolism decline in patients with Alzheimer's disease. Brain. 2021 Dec 31;144(12):3742-3755. doi: 10.1093/brain/awab222. PMID 34145880

RESULTS

PARTICIPANT FLOW:
Groups:
- Riluzole: Riluzole 50mg twice a day
- Placebo: Matching placebo twice a day
Period: Overall Study
Arm/Group | Riluzole | Placebo
Started | 26 | 24
Completed | 22 | 20
Not Completed | 4 | 4
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Riluzole | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (7.7) | 75.3 (5.8) | 74.98 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 6 | 10 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1
  Black/non-Hispanic | 1 | 0 | 1
  Latino/Hispanic | 0 | 1 | 1
  White/non-Hispanic | 19 | 20 | 39
Education [Mean (Standard Deviation); unit: years] | 15.1 (3.1) | 15.9 (3.0) | 15.5 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Imaging Biomarkers FDG-PET SUVR in Regions of Interest
Description: Change from baseline to 6 months in cerebral glucose metabolism measured with FDG PET in posterior cingulate cortex, hippocampus, precuneus, and medial temporal, lateral temporal, inferior parietal, and frontal lobes, referred to collectively as our pre-specified regions of interest.
  Fluorodeoxyglucose (FDG)-positron emission tomography (PET) is an imaging procedure that measures glucose metabolism in the brain.It is a well-established Alzheimer's disease biomarker and predictor of disease progression. For each FDG PET scan, 5 mCi of fluorodeoxyglucose was administered followed by a 40 minute uptake period during which the participant was in a resting state. Images were acquired on a Siemens Biograph 64mCT scanner as a series of 4 frames of 5 minutes each. Using SPM12 (Wellcome Trust), motion correction was performed and frames averaged into a static image. Each 6 month scan was coregistered to the baseline FDG scan, which was co-registered to the participant's T1-weighted MRI scan.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: Standardized Uptake Value Ratios (SUVRs)
Arm/Group | Placebo | Riluzole
Number analyzed (Participants) | 20 | 22
Standardized Uptake Value Ratios (SUVRs)
  Posterior cingulate | -0.048 (0.035) | -0.005 (0.035)
  Precuneus | -0.032 (0.028) | -0.007 (0.032)
  Temporal | -0.023 (0.033) | 0.002 (0.029)
  Frontal | -0.129 (0.066) | -0.077 (0.072)
  Parietal | -0.020 (0.027) | -0.005 (0.024)
  Hippocampus | -0.018 (0.034) | -0.002 (0.029)
  Right Hippocampus | -0.021 (0.036) | 0.002 (0.027)
  AD Progression score | 0.579 (0.607) | 0.245 (0.558)
  Post Cing - Precuneus | -0.041 (0.042) | -0.006 (0.038)
  Orbitofrontal | -0.019 (0.044) | 0.014 (0.036)

2. Primary Outcome: Imaging Biomarkers N-acetylaspartate (NAA) in Posterior Cingulate (PC) Measured Through 1H MRS
Description: N-acetylaspartate (NAA) is a neuronal viability marker measured through magnetic resonance spectroscopy (1H MRS).In vivo brain levels of NAA, glutamate, tCr and other major metabolites were obtained using 1H MRS and a 2x2x2-cm3 Posterior Cingulate Cortex (PC) voxel of interest in approximately 6.5 minutes using the constant-time point-resolved spectroscopy (CT-PRESS) technique with TE 30 ms, 129 constant-time increments (t1) of 0.8ms, and TR 1500 ms and a receive-only 8-channel phased-array head coil.The levels of NAA and other metabolites were expressed semi-quantitatively as ratios of peak areas relative to that of the unsuppressed water signal (W) from the same voxels. For consistency with earlier MRS literature, levels of the same metabolites were also expressed as peak ratios relative to tCr area in the same voxel.
Time Frame: Changes from baseline to 6 months
Population: Some participants could not complete MRS study due to multiple reasons (eg could not tolerate lengthy exam, did not return to visit etc) or did complete it but quality control of the MRS spectra did not pass screening criteria for analysis.
Measure: Mean (Standard Deviation); unit: Ratios
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 19 | 19
Ratios
  BASELINE (NAA/W) | 0.3843874 (0.0815156) | 0.4274546 (0.0684472)
  3 MONTHS (NAA/W): number analyzed (Participants) | 19 | 18
  3 MONTHS (NAA/W) | 0.3996655 (0.0927727) | 0.4248429 (0.0774599)
  6 MONTHS (NAA/W): number analyzed (Participants) | 17 | 18
  6 MONTHS (NAA/W) | 0.3784181 (0.0758756) | 0.4415926 (0.1039630)
  BASELINE (NAA/tCr) | 1.4488809 (0.1731644) | 1.4802620 (0.1412636)
  3 MONTHS (NAA/tCr): number analyzed (Participants) | 19 | 18
  3 MONTHS (NAA/tCr) | 1.4271889 (0.1140340) | 1.4766125 (0.1304353)
  6 MONTHS (NAA/tCr): number analyzed (Participants) | 17 | 18
  6 MONTHS (NAA/tCr) | 1.4594796 (0.1458860) | 1.4811814 (0.1474927)

3. Secondary Outcome: Glutamate Levels Measured Through 1H MRS
Description: In vivo measurement of glutamate with 1H magnetic resonance spectroscopy (MRS) (a neuroimaging study) in posterior cingulate as a marker of target engagement at three and six months compared to baseline.In vivo brain levels of glutamate, tCr and other major metabolites were obtained using 1H MRS and a 2x2x2-cm3 Posterior Cingulate Cortex voxel of interest in approximately 6.5 minutes using the constant-time point-resolved spectroscopy (CT-PRESS) technique with TE 30 ms, 129 constant-time increments (t1) of 0.8ms, and TR 1500 ms and a receive-only 8-channel phased-array head coil.The levels of glutamate and other metabolites were expressed semi-quantitatively as ratios of peak areas relative to that of the unsuppressed water signal (W) from the same voxels. For consistency with earlier MRS literature, levels of the same metabolites were also expressed as peak ratios relative to tCr area in the same voxel.
Time Frame: Change from baseline to 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratios
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 19 | 19
Ratios
  BASELINE (Glu/W) | 0.0598059 (0.0164069) | 0.0677906 (0.0133271)
  3 MONTHS (Glu/W): number analyzed (Participants) | 19 | 18
  3 MONTHS (Glu/W) | 0.0579899 (0.0181040) | 0.0646162 (0.0107094)
  6 MONTHS (Glu/W): number analyzed (Participants) | 17 | 18
  6 MONTHS (Glu/W) | 0.0609985 (0.0156960) | 0.0633453 (0.0147764)
  BASELINE (Glu/tCr) | 0.2280186 (0.0543718) | 0.2367567 (0.0484442)
  3 MONTHS (Glu/tCr): number analyzed (Participants) | 19 | 18
  3 MONTHS (Glu/tCr) | 0.2080647 (0.0515160) | 0.2285644 (0.0441709)
  6 MONTHS (Glu/tCr): number analyzed (Participants) | 17 | 18
  6 MONTHS (Glu/tCr) | 0.2339366 (0.0370164) | 0.2162526 (0.0426140)

4. Secondary Outcome: Alzheimer's Disease Assessment Scale (ADAS) - Cognitive Subscale (ADAScog)
Description: The ADAS comprises two subscales, cognitive and non-cognitive. The Cognitive Subscale (ADAScog) is a psychometric instrument that includes 11 tasks and evaluates memory, attention, reasoning, language, orientation, and praxis, scored from 0 to 70. The full ADAS total is scored by summing the number of errors made on each task on a range from 0 to 150 so that higher scores indicate worse performance.The non-cognitive component was not used in this study. Obtained for correlation with neuroimaging biomarkers.
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 20
score on a scale
  BASELINE | 22.4981818 (7.8875264) | 17.9005000 (7.4614719)
  6 MONTHS | 21.8022727 (9.7334313) | 18.8495000 (9.2608983)

5. Secondary Outcome: Neuropsychiatry Inventory - NPI
Description: NPI assesses psychopathology in participants with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with the participant's behavior. Total score ranges from 0 to 144; Higher scores indicate greater disease severity.
  Obtained for correlation with neuroimaging
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 20
score on a scale
  BASELINE | 9.6363636 (9.1627894) | 10.2000000 (11.1383642)
  6 MONTHS | 9.0909091 (6.6254135) | 14.0500000 (12.8082005)

6. Secondary Outcome: ADCS Activities of Daily Living
Description: ADCS-ADL is a 23-item inventory developed as a Rater-administered questionnaire answered by the participant's caregiver. It measures performance of basic and instrumental activities of daily living by participants. The total score ranges from 0 to 78, with lower scores indicating greater disease severity.
  Obtained for correlation with neuroimaging
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 22 | 20
score on a scale
  BASELINE | 68.3636364 (9.5096215) | 68.0500000 (9.3215935)
  6 MONTHS | 65.5000000 (11.5377228) | 64.3000000 (10.7757037)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Riluzole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/26 | 1/24
Other Adverse Events (participants affected / at risk) | 21/26 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=26) | Placebo (N=24)
GI (Gastrointestinal disorders) | 1 (1) | 0 (0) — Gastrointestinal hemorrhage with hospitalization and study article discontinuation
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — laboratory abnormalities (thrombocytopenia) with study article discontinuation
Cardiac (Cardiac disorders) | 0 (0) | 1 (1) — bradycardia and pacemaker placement with study article discontinuation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riluzole (N=26) | Placebo (N=24)
Abdominal discomfort (Gastrointestinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dizziness (General disorders) | 4 | 1
Urinary frequency (Renal and urinary disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Elevated liver enzymes (Hepatobiliary disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 4
Paranoia (Psychiatric disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Fatigue (General disorders) | 1 | 2
Somnolence (General disorders) | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
1.Sample size was relatively small, and results require replication in larger-sample studies. 2.lack of amyloid characterization. 3.MRS is unable to differentiate neurotransmitter or vesicular and metabolic pools of glutamate. Longitudinal MRS measurements can be subject to technical variability and head motion. 4. the study was not powered for neuropsychological outcome and clinical changes must be viewed only as directional/exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT01703117/Prot_SAP_000.pdf